CLINICAL TRIAL: NCT03000322
Title: Investigation of a Cooling Vest in Men With Chemotherapy-Induced Hot Flashes
Brief Title: Cooling Vest in Men With Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-16-680
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes

ARMS (1):
- Cooling Vest (Experimental): During the four-week Treatment Period, participants should use the Cooling Vest two times per day (once in the morning for one hour and once in the evening for one hour.)
  Interventions: Device: Cooling Vest

INTERVENTIONS:
Device: Cooling Vest — A cool therapy device intended to provide moderate, controlled cooling (approximately 15C/59F) by absorbing heat. The material in the vest is safe, non-toxic, and eco-friendly.

SUMMARY:
This study is intended to determine the efficacy of the Cooling Vest in reducing the frequency and intensity of hot flashes and night sweats in men undergoing chemotherapy treatment for prostate cancer.

DETAILED DESCRIPTION:
The Cooling Vest is a vest manufactured by Nanohealth, Inc. It is a cool therapy device intended to provide moderate, controlled cooling (approximately 15C/59F) by absorbing heat. The material in the vest is safe, non-toxic, and eco-friendly.

This study attempts to collect data on the effects of the Cooling Vest in men with hot flashes and night sweats due to the side effects of chemotherapy. Participants will use the vest for 4 weeks and questionnaires will be used to determine effect.

ELIGIBILITY:
Inclusion Criteria:

* Males, who are at least 18 years old.
* Self-reports having at least two (2) daily hot flashes associated with prostate cancer chemotherapy-induced hot flashes and night sweats.

Exclusion Criteria:

* Has another existing medical condition that would prevent study compliance.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
change in number of daily hot flashes | 4 weeks
  diary will be used to record the number of daily hot flashes
change in the intensity of daily hot flashes | 4 weeks
  diary will be used to record the severity of daily hot flashes

CONTACTS AND LOCATIONS:
Overall Officials: Eric Margolis, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Urology Center Research Institute, Englewood, New Jersey, United States